CLINICAL TRIAL: NCT03023384
Title: Feasibility Study of the Use of Intermediate Doses of Cytarabine Associated With Autologous Hematopoietic Stem Cells as Consolidation Treatment of Young Adults With Low- or Intermediate-risk de Novo Acute Myeloid Leukemia
Brief Title: Feasibility Study of Intermediate Doses of ARA-C With Autologous SCT as Consolidation of Low/Intermediate-risk AML
Acronym: ICAML2015
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Consortium on Acute Leukemias (Other)
Responsible Party: Sponsor
Other Study IDs: ICAML2015
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Chemotherapy; Autologous Stem Cell Transplantation; Developing country; Clinical network
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood and Bone Marrow Aspirate
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Create a network of institutions in developing countries that will perform AML diagnosis, risk classification, treatment, supportive care and follow-up evaluation according to a common protocol and will register data using common clinical research forms (CRFs) in a single database and available on the internet.

DETAILED DESCRIPTION:
1. Compare overall survival and disease-free survival of patients with acute myeloid leukemia classified according the European LeukemiaNet treated in participating South American hospitals with the results reported in developed countries.
2. Compare overall survival and disease-free survival of patients with AML low or intermediate risk treated with two cycles of cytarabine in intermediate dose versus one cytarabine cycle at the same dose followed by autologous SCT as consolidation. The risk will be established according to the classification of the European LeukemiaNet.
3. Create a network of institutions in developing countries that will perform AML diagnosis, risk classification, treatment, supportive care and follow-up evaluation according to a common protocol and will register data using common clinical research forms (CRFs) in a single database and available on the internet
4. Using National Reference Laboratories, provide cytogenetic and molecular methods for all institutions participating in the network, thus allowing rapid diagnosis and risk stratification of AML cases according to the European LeukemiaNet structure;
5. Develop a method of assessing minimal residual disease based on flow cytometry adapted to local resources and capable of guiding therapeutic decisions;
6. Determine the time interval between: a) diagnosis and risk group determination; b) the first cycle of consolidation chemotherapy and autologous hematopoietic stem cells infusion;
7. Determine the frequency and etiologic agent of infections associated with treatment, the number and average duration of hospitalization due to episodes of neutropenia;
8. Create a bank of samples of bone marrow from AML patients at different times of treatment;
9. Determine the disease-free survival and the cumulative incidence rate of relapse and non-relapse mortality and compare them between chemotherapy alone and chemotherapy plus autologous SCT cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myeloid leukemia (AML) diagnosis according to WHO criteria;
2. AML not treated previously, including: de novo AML or secondary to myelodysplastic syndromes;
3. Absence of t(15;17), or PML-RARA rearrangement and its variants (acute promyelocytic leukemia diagnosis);
4. Age greater than or equal to 18 years old or lower than or equal to 65 years old;
5. Functional status ECOG from 0 to 2;
6. Signed informed consent;
7. Ability to follow the protocol procedures;
8. Willingness to use birth control methods during the treatment until its conclusion;
9. Adequate renal and liver function:

   * Bilirubin ≤ 1.5x the upper limit of normality;
   * AST and ALT ≤ 2.5x the upper limit of normality;
   * Creatinine ≤ 2.5 mg/dL.
10. Suitable cardiac function: left ventricular ejection fraction ≥ 50%.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL) diagnosis according to WHO criteria;
2. Diagnosis of acute leukemia of ambiguous lineage, biphenotypic acute leukemia or undifferentiated acute leukemia, according to WHO criteria;
3. AML previously treated, except with hydroxyurea administration for cytoreduction;
4. Age greater than 65 years old or lower than 18 years old;
5. Functional status ECOG greater than 2;
6. Do not sign the informed consent;
7. Inability to follow the protocol procedures;
8. Be fertile female who are unwilling to take any birth control method during the treatment;
9. Hypersensitivity to any drug of the treatment protocol;
10. Positive serology for HIV;
11. Altered liver and renal function not related to the primary disease (AML):

    * Bilirubin > 1.5x the upper limit of normality
    * AST and ALT > the 2.5x upper limit of normality
    * Creatinine > 2.5 mg/dL

n) Altered cardiac function, with LVEF <50%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Acute Myeloid Leukemia
Sampling Method: Probability Sample
Enrollment: 547 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 years
  Time from diagnosis until relapse

SECONDARY OUTCOMES:
Overall survival | 2 years
  Time from diagnosis until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo M Rego, MD, Principal Investigator — University of Sao Paulo
Locations (6):
- Brazil (6):
  - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Unicamp, Campinas, São Paulo
  - Hospital das Clinicas de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital Mario Covas, Santo André, São Paulo
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burnett A, Wetzler M, Lowenberg B. Therapeutic advances in acute myeloid leukemia. J Clin Oncol. 2011 Feb 10;29(5):487-94. doi: 10.1200/JCO.2010.30.1820. Epub 2011 Jan 10. PMID 21220605
- [Background] Lowenberg B, Downing JR, Burnett A. Acute myeloid leukemia. N Engl J Med. 1999 Sep 30;341(14):1051-62. doi: 10.1056/NEJM199909303411407. No abstract available. PMID 10502596
- [Background] Lowenberg B. Sense and nonsense of high-dose cytarabine for acute myeloid leukemia. Blood. 2013 Jan 3;121(1):26-8. doi: 10.1182/blood-2012-07-444851. PMID 23287624
- [Background] Lowenberg B, Pabst T, Vellenga E, van Putten W, Schouten HC, Graux C, Ferrant A, Sonneveld P, Biemond BJ, Gratwohl A, de Greef GE, Verdonck LF, Schaafsma MR, Gregor M, Theobald M, Schanz U, Maertens J, Ossenkoppele GJ; Dutch-Belgian Cooperative Trial Group for Hemato-Oncology (HOVON) and Swiss Group for Clinical Cancer Research (SAKK) Collaborative Group. Cytarabine dose for acute myeloid leukemia. N Engl J Med. 2011 Mar 17;364(11):1027-36. doi: 10.1056/NEJMoa1010222. PMID 21410371
- [Background] Mrozek K, Marcucci G, Nicolet D, Maharry KS, Becker H, Whitman SP, Metzeler KH, Schwind S, Wu YZ, Kohlschmidt J, Pettenati MJ, Heerema NA, Block AW, Patil SR, Baer MR, Kolitz JE, Moore JO, Carroll AJ, Stone RM, Larson RA, Bloomfield CD. Prognostic significance of the European LeukemiaNet standardized system for reporting cytogenetic and molecular alterations in adults with acute myeloid leukemia. J Clin Oncol. 2012 Dec 20;30(36):4515-23. doi: 10.1200/JCO.2012.43.4738. Epub 2012 Sep 17. PMID 22987078
- [Background] Buchner T, Schlenk RF, Schaich M, Dohner K, Krahl R, Krauter J, Heil G, Krug U, Sauerland MC, Heinecke A, Spath D, Kramer M, Scholl S, Berdel WE, Hiddemann W, Hoelzer D, Hehlmann R, Hasford J, Hoffmann VS, Dohner H, Ehninger G, Ganser A, Niederwieser DW, Pfirrmann M. Acute Myeloid Leukemia (AML): different treatment strategies versus a common standard arm--combined prospective analysis by the German AML Intergroup. J Clin Oncol. 2012 Oct 10;30(29):3604-10. doi: 10.1200/JCO.2012.42.2907. Epub 2012 Sep 10. PMID 22965967
- [Background] Pfirrmann M, Ehninger G, Thiede C, Bornhauser M, Kramer M, Rollig C, Hasford J, Schaich M; Study Alliance Leukaemia (SAL). Prediction of post-remission survival in acute myeloid leukaemia: a post-hoc analysis of the AML96 trial. Lancet Oncol. 2012 Feb;13(2):207-14. doi: 10.1016/S1470-2045(11)70326-6. Epub 2011 Dec 22. PMID 22197676
- [Background] Grimwade D. The changing paradigm of prognostic factors in acute myeloid leukaemia. Best Pract Res Clin Haematol. 2012 Dec;25(4):419-25. doi: 10.1016/j.beha.2012.10.004. Epub 2012 Nov 4. PMID 23200538
- [Background] Dohner H, Estey EH, Amadori S, Appelbaum FR, Buchner T, Burnett AK, Dombret H, Fenaux P, Grimwade D, Larson RA, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz MA, Sierra J, Tallman MS, Lowenberg B, Bloomfield CD; European LeukemiaNet. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood. 2010 Jan 21;115(3):453-74. doi: 10.1182/blood-2009-07-235358. Epub 2009 Oct 30. PMID 19880497
- [Background] Rollig C, Bornhauser M, Thiede C, Taube F, Kramer M, Mohr B, Aulitzky W, Bodenstein H, Tischler HJ, Stuhlmann R, Schuler U, Stolzel F, von Bonin M, Wandt H, Schafer-Eckart K, Schaich M, Ehninger G. Long-term prognosis of acute myeloid leukemia according to the new genetic risk classification of the European LeukemiaNet recommendations: evaluation of the proposed reporting system. J Clin Oncol. 2011 Jul 10;29(20):2758-65. doi: 10.1200/JCO.2010.32.8500. Epub 2011 May 31. PMID 21632498
- [Background] Burnett AK, Wheatley K, Goldstone AH, Stevens RF, Hann IM, Rees JH, Harrison G; Medical Research Council Adult and Paediatric Working Parties. The value of allogeneic bone marrow transplant in patients with acute myeloid leukaemia at differing risk of relapse: results of the UK MRC AML 10 trial. Br J Haematol. 2002 Aug;118(2):385-400. doi: 10.1046/j.1365-2141.2002.03724.x. PMID 12139722
- [Background] Koreth J, Schlenk R, Kopecky KJ, Honda S, Sierra J, Djulbegovic BJ, Wadleigh M, DeAngelo DJ, Stone RM, Sakamaki H, Appelbaum FR, Dohner H, Antin JH, Soiffer RJ, Cutler C. Allogeneic stem cell transplantation for acute myeloid leukemia in first complete remission: systematic review and meta-analysis of prospective clinical trials. JAMA. 2009 Jun 10;301(22):2349-61. doi: 10.1001/jama.2009.813. PMID 19509382
- [Background] Majhail NS, Bajorunaite R, Lazarus HM, Wang Z, Klein JP, Zhang MJ, Rizzo JD. High probability of long-term survival in 2-year survivors of autologous hematopoietic cell transplantation for AML in first or second CR. Bone Marrow Transplant. 2011 Mar;46(3):385-92. doi: 10.1038/bmt.2010.115. Epub 2010 May 17. PMID 20479710
- [Background] Nakasone H, Izutsu K, Wakita S, Yamaguchi H, Muramatsu-Kida M, Usuki K. Autologous stem cell transplantation with PCR-negative graft would be associated with a favorable outcome in core-binding factor acute myeloid leukemia. Biol Blood Marrow Transplant. 2008 Nov;14(11):1262-9. doi: 10.1016/j.bbmt.2008.08.012. PMID 18940681
- [Background] Breems DA, Boogaerts MA, Dekker AW, Van Putten WL, Sonneveld P, Huijgens PC, Van der Lelie J, Vellenga E, Gratwohl A, Verhoef GE, Verdonck LF, Lowenberg B. Autologous bone marrow transplantation as consolidation therapy in the treatment of adult patients under 60 years with acute myeloid leukaemia in first complete remission: a prospective randomized Dutch-Belgian Haemato-Oncology Co-operative Group (HOVON) and Swiss Group for Clinical Cancer Research (SAKK) trial. Br J Haematol. 2005 Jan;128(1):59-65. doi: 10.1111/j.1365-2141.2004.05282.x. PMID 15606550
- [Background] Wang J, Ouyang J, Zhou R, Chen B, Yang Y. Autologous hematopoietic stem cell transplantation for acute myeloid leukemia in first complete remission: a meta-analysis of randomized trials. Acta Haematol. 2010;124(2):61-71. doi: 10.1159/000314273. Epub 2010 Jul 10. PMID 20616541
- [Background] Nucci M, Garnica M, Gloria AB, Lehugeur DS, Dias VC, Palma LC, Cappellano P, Fertrin KY, Carlesse F, Simoes B, Bergamasco MD, Cunha CA, Seber A, Ribeiro MP, Queiroz-Telles F, Lee ML, Chauffaille ML, Silla L, de Souza CA, Colombo AL. Invasive fungal diseases in haematopoietic cell transplant recipients and in patients with acute myeloid leukaemia or myelodysplasia in Brazil. Clin Microbiol Infect. 2013 Aug;19(8):745-51. doi: 10.1111/1469-0691.12002. Epub 2012 Sep 25. PMID 23009319
- [Background] Levi I, Grotto I, Yerushalmi R, Ben-Bassat I, Shpilberg O. Meta-analysis of autologous bone marrow transplantation versus chemotherapy in adult patients with acute myeloid leukemia in first remission. Leuk Res. 2004 Jun;28(6):605-12. doi: 10.1016/j.leukres.2003.10.029. PMID 15120937
- [Background] Zittoun RA, Mandelli F, Willemze R, de Witte T, Labar B, Resegotti L, Leoni F, Damasio E, Visani G, Papa G, et al. Autologous or allogeneic bone marrow transplantation compared with intensive chemotherapy in acute myelogenous leukemia. European Organization for Research and Treatment of Cancer (EORTC) and the Gruppo Italiano Malattie Ematologiche Maligne dell'Adulto (GIMEMA) Leukemia Cooperative Groups. N Engl J Med. 1995 Jan 26;332(4):217-23. doi: 10.1056/NEJM199501263320403. PMID 7808487
- [Background] Keating A, DaSilva G, Perez WS, Gupta V, Cutler CS, Ballen KK, Cairo MS, Camitta BM, Champlin RE, Gajewski JL, Lazarus HM, Lill M, Marks DI, Nabhan C, Schiller GJ, Socie G, Szer J, Tallman MS, Weisdorf DJ. Autologous blood cell transplantation versus HLA-identical sibling transplantation for acute myeloid leukemia in first complete remission: a registry study from the Center for International Blood and Marrow Transplantation Research. Haematologica. 2013 Feb;98(2):185-92. doi: 10.3324/haematol.2012.062059. Epub 2012 Sep 14. PMID 22983587
- [Background] Capra M, Vilella L, Pereira WV, Coser VM, Fernandes MS, Schilling MA, Almeida D, Gross M, Leite M, Hellwig T, Natchigal G, Zelmanowicz A, Paskulin G, Neumann J, Silla L. Estimated number of cases, regional distribution and survival of patients diagnosed with acute myeloid leukemia between 1996 and 2000 in Rio Grande do Sul, Brazil. Leuk Lymphoma. 2007 Dec;48(12):2381-6. doi: 10.1080/10428190701713622. PMID 18067014
- [Background] Chan LL, Abdel-Latif ME, Ariffin WA, Ariffin H, Lin HP. Treating childhood acute myeloid leukaemia with the AML-BFM-83 protocol: experience in a developing country. Br J Haematol. 2004 Sep;126(6):799-805. doi: 10.1111/j.1365-2141.2004.05129.x. PMID 15352983
- [Background] Eid KA, Miranda EC, Vigorito AC, Aranha FJ, Oliveira GB, De Souza CA. The availability of full match sibling donors and feasibility of allogeneic bone marrow transplantation in Brazil. Braz J Med Biol Res. 2003 Mar;36(3):315-21. doi: 10.1590/s0100-879x2003000300005. Epub 2003 Mar 7. PMID 12640495
- [Background] Giebel S, Labopin M, Ehninger G, Beelen D, Blaise D, Ganser A, Bacigalupo A, Czerw T, Holowiecki J, Fagundes EM, Nowara E, Frassoni F, Rocha V; Acute Leukemia Working Party of the European Group for Blood and Marrow Transplantation. Association of Human Development Index with rates and outcomes of hematopoietic stem cell transplantation for patients with acute leukemia. Blood. 2010 Jul 8;116(1):122-8. doi: 10.1182/blood-2010-01-266478. Epub 2010 Apr 15. PMID 20395416
- [Background] Howard SC, Ortiz R, Baez LF, Cabanas R, Barrantes J, Fu L, Pena A, Samudio A, Vizcaino M, Rodriguez-Galindo C, Barr RD, Conter V, Biondi A, Masera G; MISPHO Consortium Writing Committee. Protocol-based treatment for children with cancer in low income countries in Latin America: a report on the recent meetings of the Monza International School of Pediatric Hematology/Oncology (MISPHO)--part II. Pediatr Blood Cancer. 2007 Apr;48(4):486-90. doi: 10.1002/pbc.20989. PMID 16883600
- [Background] Sandes AF, Ribeiro JC, Barroso RS, Silva MR, Chauffaille ML. Improving the outcomes of elderly patients with acute myeloid leukemia in a Brazilian University Hospital. Clinics (Sao Paulo). 2011;66(8):1335-40. doi: 10.1590/s1807-59322011000800005. PMID 21915480
- [Background] Xu XJ, Tang YM, Song H, Yang SL, Shi SW, Wei J. Long-term outcome of childhood acute myeloid leukemia in a developing country: experience from a children's hospital in China. Leuk Lymphoma. 2010 Dec;51(12):2262-9. doi: 10.3109/10428194.2010.518653. Epub 2010 Oct 7. PMID 20929322
- [Background] Rowe JM. Optimal induction and post-remission therapy for AML in first remission. Hematology Am Soc Hematol Educ Program. 2009:396-405. doi: 10.1182/asheducation-2009.1.396. PMID 20008225
- [Background] Fagundes EM, Rocha V, Gloria AB, Clementino NC, Quintao JS, Guimaraes JP, Pedroso ER, Viana MB. De novo acute myeloid leukemia in adults younger than 60 years of age: socioeconomic aspects and treatment results in a Brazilian university center. Leuk Lymphoma. 2006 Aug;47(8):1557-64. doi: 10.1080/10428190600627055. PMID 16966267
- [Background] Vardiman JW, Thiele J, Arber DA, Brunning RD, Borowitz MJ, Porwit A, Harris NL, Le Beau MM, Hellstrom-Lindberg E, Tefferi A, Bloomfield CD. The 2008 revision of the World Health Organization (WHO) classification of myeloid neoplasms and acute leukemia: rationale and important changes. Blood. 2009 Jul 30;114(5):937-51. doi: 10.1182/blood-2009-03-209262. Epub 2009 Apr 8. PMID 19357394
- [Background] Scholl C, Gilliland DG, Frohling S. Deregulation of signaling pathways in acute myeloid leukemia. Semin Oncol. 2008 Aug;35(4):336-45. doi: 10.1053/j.seminoncol.2008.04.004. PMID 18692684
- [Background] Sternberg DW, Gilliland DG. The role of signal transducer and activator of transcription factors in leukemogenesis. J Clin Oncol. 2004 Jan 15;22(2):361-71. doi: 10.1200/JCO.2004.10.124. PMID 14722044
- [Background] Lin HK, Bergmann S, Pandolfi PP. Deregulated TGF-beta signaling in leukemogenesis. Oncogene. 2005 Aug 29;24(37):5693-700. doi: 10.1038/sj.onc.1208923. PMID 16123802
- [Background] Moe-Behrens GH, Pandolfi PP. Targeting aberrant transcriptional repression in acute myeloid leukemia. Rev Clin Exp Hematol. 2003 Jun;7(2):139-59. PMID 14763160
- [Background] Kosmider O, Moreau-Gachelin F. From mice to human: the "two-hit model" of leukemogenesis. Cell Cycle. 2006 Mar;5(6):569-70. doi: 10.4161/cc.5.6.2577. Epub 2006 Mar 15. No abstract available. PMID 16582609
- [Background] Grimwade D, Mrozek K. Diagnostic and prognostic value of cytogenetics in acute myeloid leukemia. Hematol Oncol Clin North Am. 2011 Dec;25(6):1135-61, vii. doi: 10.1016/j.hoc.2011.09.018. PMID 22093581
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Ohtake S, Miyawaki S, Fujita H, Kiyoi H, Shinagawa K, Usui N, Okumura H, Miyamura K, Nakaseko C, Miyazaki Y, Fujieda A, Nagai T, Yamane T, Taniwaki M, Takahashi M, Yagasaki F, Kimura Y, Asou N, Sakamaki H, Handa H, Honda S, Ohnishi K, Naoe T, Ohno R. Randomized study of induction therapy comparing standard-dose idarubicin with high-dose daunorubicin in adult patients with previously untreated acute myeloid leukemia: the JALSG AML201 Study. Blood. 2011 Feb 24;117(8):2358-65. doi: 10.1182/blood-2010-03-273243. Epub 2010 Aug 6. PMID 20693429
- [Background] Teuffel O, Leibundgut K, Lehrnbecher T, Alonzo TA, Beyene J, Sung L. Anthracyclines during induction therapy in acute myeloid leukaemia: a systematic review and meta-analysis. Br J Haematol. 2013 Apr;161(2):192-203. doi: 10.1111/bjh.12233. Epub 2013 Feb 8. PMID 23398482
- [Background] Burnett AK. New induction and postinduction strategies in acute myeloid leukemia. Curr Opin Hematol. 2012 Mar;19(2):76-81. doi: 10.1097/MOH.0b013e3283500a92. PMID 22248879
- [Background] Rego EM, Jacomo RH. Epidemiology and treatment of acute promyelocytic leukemia in latin america. Mediterr J Hematol Infect Dis. 2011;3(1):e2011049. doi: 10.4084/MJHID.2011.049. Epub 2011 Oct 24. PMID 22110899
- [Background] Rego EM, Kim HT, Ruiz-Arguelles GJ, Undurraga MS, Uriarte Mdel R, Jacomo RH, Gutierrez-Aguirre H, Melo RA, Bittencourt R, Pasquini R, Pagnano K, Fagundes EM, Chauffaille Mde L, Chiattone CS, Martinez L, Meillon LA, Gomez-Almaguer D, Kwaan HC, Garces-Eisele J, Gallagher R, Niemeyer CM, Schrier SL, Tallman M, Grimwade D, Ganser A, Berliner N, Ribeiro RC, Lo-Coco F, Lowenberg B, Sanz MA. Improving acute promyelocytic leukemia (APL) outcome in developing countries through networking, results of the International Consortium on APL. Blood. 2013 Mar 14;121(11):1935-43. doi: 10.1182/blood-2012-08-449918. Epub 2013 Jan 14. PMID 23319575
- [Background] Bucaneve G, Micozzi A, Menichetti F, Martino P, Dionisi MS, Martinelli G, Allione B, D'Antonio D, Buelli M, Nosari AM, Cilloni D, Zuffa E, Cantaffa R, Specchia G, Amadori S, Fabbiano F, Deliliers GL, Lauria F, Foa R, Del Favero A; Gruppo Italiano Malattie Ematologiche dell'Adulto (GIMEMA) Infection Program. Levofloxacin to prevent bacterial infection in patients with cancer and neutropenia. N Engl J Med. 2005 Sep 8;353(10):977-87. doi: 10.1056/NEJMoa044097. PMID 16148283
- [Background] Gafter-Gvili A, Fraser A, Paul M, Vidal L, Lawrie TA, van de Wetering MD, Kremer LC, Leibovici L. Antibiotic prophylaxis for bacterial infections in afebrile neutropenic patients following chemotherapy. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD004386. doi: 10.1002/14651858.CD004386.pub3. PMID 22258955
- [Background] Robenshtok E, Gafter-Gvili A, Goldberg E, Weinberger M, Yeshurun M, Leibovici L, Paul M. Antifungal prophylaxis in cancer patients after chemotherapy or hematopoietic stem-cell transplantation: systematic review and meta-analysis. J Clin Oncol. 2007 Dec 1;25(34):5471-89. doi: 10.1200/JCO.2007.12.3851. Epub 2007 Oct 1. PMID 17909198
- [Background] Gafter-Gvili A, Fraser A, Paul M, Leibovici L. Meta-analysis: antibiotic prophylaxis reduces mortality in neutropenic patients. Ann Intern Med. 2005 Jun 21;142(12 Pt 1):979-95. doi: 10.7326/0003-4819-142-12_part_1-200506210-00008. PMID 15968013
- [Background] Garnica M, Nouer SA, Pellegrino FL, Moreira BM, Maiolino A, Nucci M. Ciprofloxacin prophylaxis in high risk neutropenic patients: effects on outcomes, antimicrobial therapy and resistance. BMC Infect Dis. 2013 Jul 31;13:356. doi: 10.1186/1471-2334-13-356. PMID 23899356
- [Background] Vellenga E, van Putten W, Ossenkoppele GJ, Verdonck LF, Theobald M, Cornelissen JJ, Huijgens PC, Maertens J, Gratwohl A, Schaafsma R, Schanz U, Graux C, Schouten HC, Ferrant A, Bargetzi M, Fey MF, Lowenberg B; Dutch-Belgian Hemato-Oncology Cooperative Group (HOVON); Swiss Group for Clinical Cancer Research Collaborative Group (SAKK). Autologous peripheral blood stem cell transplantation for acute myeloid leukemia. Blood. 2011 Dec 1;118(23):6037-42. doi: 10.1182/blood-2011-07-370247. Epub 2011 Sep 27. PMID 21951683
- [Background] Klein JP, Andersen PK. Regression modeling of competing risks data based on pseudovalues of the cumulative incidence function. Biometrics. 2005 Mar;61(1):223-9. doi: 10.1111/j.0006-341X.2005.031209.x. PMID 15737097